CLINICAL TRIAL: NCT01778634
Title: A Phase IIb Randomized, Placebo-controlled, Double-blind Trial of Azithromycin to Eradicate Ureaplasma Respiratory Tract Infection in Preterm Infants
Brief Title: Trial of Intravenous Azithromycin to Eradicate Ureaplasma Respiratory Tract Infection in Preterm Infants
Acronym: AZIPIII
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Mercy Medical Center (Other); Johns Hopkins University (Other); University of Virginia (Other); University of Alabama at Birmingham (Other); Christiana Care Health Services (Other)
Responsible Party: Principal Investigator, Rose Viscardi, Professor of Pediatrics, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HP-00054998; R01HD067126 (NIH)
Record Dates: First submitted 2013-01-22; First posted 2013-01-29 (Estimated); Results first posted 2018-05-17 (Actual); Last update posted 2020-11-30 (Actual); Status verified 2020-11

CONDITIONS: Ureaplasma Infections
Keywords: Ureaplasma parvum; Ureaplasma urealyticum; prematurity; bronchopulmonary dysplasia; azithromycin
MeSH Terms: conditions — Ureaplasma Infections; Premature Birth; Bronchopulmonary Dysplasia | interventions — Azithromycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (5% dextrose) (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- Azithromycin (Experimental): Azithromycin intravenous (2 mg/ml) 20 mg/kg every 24h x 3 days
  Interventions: Drug: Azithromycin

INTERVENTIONS:
Drug: Azithromycin — Azithromycin intravenous 20 mg/kg every 24 h x 3 days
  Other Names: Zithromax
  Arms: Azithromycin
Drug: Placebo — D5W
  Other Names: equal volume of 5% dextrose water
  Arms: Placebo (5% dextrose)

SUMMARY:
The purpose of this study is to determine whether intravenous azithromycin is effective in eradicating Ureaplasma respiratory tract infection in preterm infants born at 24 to 28 weeks gestation.

DETAILED DESCRIPTION:
The study design will be a double-blind, placebo-controlled clinical trial to test the efficacy and safety of azithromycin 20 mg/kg x 3 days to eradicate Ureaplasma spp from the respiratory tract of preterm infants 24 weeks 0 days to 28 weeks 6 days gestation exposed to positive pressure ventilation. The primary outcome will be survival with microbiological eradication of Ureaplasma defined as survival to discharge or transfer with 3 negative cultures obtained post-therapy. Secondary outcomes will include physiologic BPD at 36 weeks post-menstrual age (PMA), overall mortality, incidence of co-morbidities of prematurity such as intraventricular hemorrhage, periventricular leukomalacia, necrotizing enterocolitis, bacterial and fungal nosocomial infection, pulmonary air leak, patent ductus arteriosus, retinopathy of prematurity, number of days of positive pressure ventilation, number of days of oxygen supplementation, use of postnatal steroids, and use of non-study antibiotics. At 6 and 18 months adjusted age, a pulmonary outcome questionnaire will be administered by phone or in person interview. At 18-22 months adjusted age, neurodevelopmental outcomes will be assessed by 1) Bayley Scale of Infant and Toddler Development, 3rd edition (BSID-III); 2) Amiel-Tison neurologic examination; 3) Gross Motor Function Classification System; and 4) medical record review for hearing impairment with or without amplification and vision impairment (vision <20/200).

ELIGIBILITY:
Inclusion Criteria:

* Gestational age 24 weeks 0 days-28weeks 6 days by best obstetrical estimate
* <72 h age
* Positive pressure ventilation for at least 1 hour duration during the first 72 hours of life
* Presence of indwelling intravenous line for drug administration

Exclusion Criteria:

* Any patient judged to be non-viable or for whom withdrawal of life support is planned
* Patients with major lethal congenital anomalies
* Triplets or higher order multiples
* Patients delivered for maternal indications (low risk of Ureaplasma colonization)
* Patients with EKG QT interval corrected for heart rate (Qtc) ≥ 450 ms
* Patients with significant hepatic impairment (direct bilirubin >1.5 mg/dL)
* Patients exposed to other systemic macrolide
* Patients with clinically suspected Ureaplasma central nervous system (CNS) infection or other confirmed bacterial/viral infection
* Patients participating in other clinical trials involving investigational products.

Ages: 2 Hours to 72 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 121 (Actual)
Dates: Start 2013-07; Primary Completion 2016-12 (Actual); Study Completion 2020-11-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rose M Viscardi, M.D., Study Chair — University of Maryland, College Park; Pamela Donohue, ScD, Principal Investigator — Johns Hopkins University; Namasivayam Ambalavanan, M.D., Principal Investigator — University of Alabama at Birmingham; David A Kaufman, M.D., Principal Investigator — University of Virginia; Michael L Terrin, M.D., Principal Investigator — University of Maryland, College Park; Susan J Dulkerian, M.D., Principal Investigator — Mercy Medical Center
Locations (7):
- United States (7):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Christiana Care Health Services, Newark, Delaware
  - University of Maryland School of Medicine, Baltimore, Maryland
  - Mercy Medical Center, Baltimore, Maryland
  - Johns Hopkins University, Baltimore, Maryland
  - Monroe Carell Jr. Children's Hospital at Vanderbilt, Nashville, Tennessee
  - University of Virginia, Charlottesville, Virginia

REFERENCES:
- [Background] Hassan HE, Othman AA, Eddington ND, Duffy L, Xiao L, Waites KB, Kaufman DA, Fairchild KD, Terrin ML, Viscardi RM. Pharmacokinetics, safety, and biologic effects of azithromycin in extremely preterm infants at risk for ureaplasma colonization and bronchopulmonary dysplasia. J Clin Pharmacol. 2011 Sep;51(9):1264-75. doi: 10.1177/0091270010382021. Epub 2010 Nov 23. PMID 21098694
- [Derived] Viscardi RM, Terrin ML, Magder LS, Davis NL, Dulkerian SJ, Waites KB, Ambalavanan N, Kaufman DA, Donohue P, Tuttle DJ, Weitkamp JH, Hassan HE, Eddington ND. Randomised trial of azithromycin to eradicate Ureaplasma in preterm infants. Arch Dis Child Fetal Neonatal Ed. 2020 Nov;105(6):615-622. doi: 10.1136/archdischild-2019-318122. Epub 2020 Mar 13. PMID 32170033

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period July 1, 2013- August 31, 2016 at 7 U.S. hospital Neonatal Intensive Care Units (NICUs).
Groups:
- Placebo (5% Dextrose): Placebo
  Placebo: D5W 10 ml/kg every 24 h x 3 days
Period: Overall Study
Arm/Group | Placebo (5% Dextrose) | Azithromycin
Started | 61 | 60
Completed | 61 | 60
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo (5% Dextrose) | Azithromycin | Total
Number analyzed (Participants) | 61 | 60 | 121
Age, Continuous [Mean (Standard Deviation); unit: weeks gestation] — gestational age in weeks
  weeks gestation | 26.2 (1.4) | 26.2 (1.4) | 26.2 (1.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 34 | 63
  Male | 32 | 26 | 58
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 61 | 58 | 119
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 43 | 21 | 64
  White | 15 | 36 | 51
  More than one race | 2 | 3 | 5
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 61 | 60 | 121
Ureaplasma-positive [Count of Participants; unit: Participants] — Any subject who had a respiratory sample (tracheal aspirate and/or nasopharyngeal aspirate) at any time point that was positive for Ureaplasma species confirmed by culture and/or PCR was considered a Ureaplasma-positive subject.
  Participants | 25 | 19 | 44

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Survival And Transfer From NICU With Microbiological Eradication of Ureaplasma
Description: Bacterial clearance (eradication) will be defined as 3 negative cultures obtained 2 and 5 days post-third dose and 21 d of age. Survival is defined as survival at time of discharge or transfer from the neonatal intensive care unit (NICU).
Time Frame: Participants will be followed for the duration of hospital stay, an expected average of 10 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (5% Dextrose) | Azithromycin
Number analyzed (Participants) | 61 | 60
Participants | 37 | 55
Statistical Analysis 1: Comparison: Placebo (5% Dextrose) vs Azithromycin; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 7.51, 95% CI 2-sided [2.53 to 22.27]

2. Secondary Outcome: Number of Participants Who Survived Until 36 Wks Postmenstrual Age With Physiologic Defined Bronchopulmonary Dysplasia (BPD) at 36 Weeks Post Menstrual Age
Description: Number of Participants who survived until 36 wks postmenstrual age with Physiologic defined bronchopulmonary dysplasia (BPD) based on oxygen-saturation monitoring
Time Frame: 36 weeks post menstrual age (one month prior to due date)
Population: Participants who survived until assessment timepoint 36 weeks post menstrual age (1 month before due date)
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (5% Dextrose) | Azithromycin
Number analyzed (Participants) | 54 | 56
Participants | 18 | 25
Statistical Analysis 1: Comparison: Placebo (5% Dextrose) vs Azithromycin; Test type: Superiority; p = 0.28, Generalized Estimating Equations; Risk Difference (RD) = .11, 95% CI 2-sided [-0.08 to 0.29] — Generalized Estimating Equations with an identity link

3. Secondary Outcome: Number of Participants With Death or Neurodevelopmental Impairment
Description: Neurodevelopmental impairment will be assigned if any of the following are present at 22-26 months adjusted age: moderate to severe cerebral palsy, bilateral blindness, bilateral hearing impairment requiring amplification, Gross Motor Function Classification System score ≥ 2, or Bayley Scale of Infant and Toddler Development, 3rd edition (BSID-III) cognitive or motor score <70.
Time Frame: 22-26 months
Population: Participants who died prior to the 22-26 months assessment timepoint and participants who were assessed for neurodevelopmental impairments
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (5% Dextrose) | Azithromycin
Number analyzed (Participants) | 52 | 53
Participants | 17 | 25
Statistical Analysis 1: Comparison: Placebo (5% Dextrose) vs Azithromycin; Test type: Superiority — P values are based on GEE to account for twins; p = 0.11, GEE

4. Secondary Outcome: Number of Participants With Pulmonary Impairment
Description: Parent report of recurrent wheezing and/or chronic cough
Time Frame: 6-26 months
Population: All participants enrolled and randomized in the trial
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (5% Dextrose) | Azithromycin
Number analyzed (Participants) | 61 | 60
Participants | 12 | 15
Statistical Analysis 1: Comparison: Placebo (5% Dextrose) vs Azithromycin; Test type: Superiority — P values are based on GEE to account for twins. The counts provided refer to to the numbers actually observed. The analysis to determine the p value accounted for the missing 11 patients using multiple imputation; p = 0.62, GEE with multiple imputation

5. Secondary Outcome: Number of Participants Who Died
Description: Number of Participants who died from any cause
Time Frame: 22-26 months
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (5% Dextrose) | Azithromycin
Number analyzed (Participants) | 61 | 60
Participants | 6 | 5
Statistical Analysis 1: Comparison: Placebo (5% Dextrose) vs Azithromycin; Test type: Superiority; p = 1.0, Fisher Exact

6. Secondary Outcome: Duration of Positive Pressure Support
Description: Combined number of days receiving mechanical ventilation plus non-invasive modes of positive pressure support.
Time Frame: Participants will be followed for the duration of hospital stay, an expected average of 10 weeks
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Placebo (5% Dextrose) | Azithromycin
Number analyzed (Participants) | 61 | 60
days | 36 [17 to 60] | 39 [19 to 56]
Statistical Analysis 1: Comparison: Placebo (5% Dextrose) vs Azithromycin; Test type: Superiority; p = 0.88, Wilcoxon (Mann-Whitney) — To include non-survivors as bad values of this outcome we imputed a high value for the participants who died. Note, because we analyzed the data using a nonparametric test, the actual value doesn't affect the analysis, only the rank of the value

7. Secondary Outcome: Duration of Oxygen Supplementation
Description: Cumulative number of days of receipt of supplemental oxygen
Time Frame: Participants will be followed for the duration of hospital stay, an expected average of 10 weeks
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Placebo (5% Dextrose) | Azithromycin
Number analyzed (Participants) | 61 | 60
days | 68 [33 to 118] | 73 [39 to 114.5]
Statistical Analysis 1: Comparison: Placebo (5% Dextrose) vs Azithromycin; Test type: Superiority; p = 0.94, Wilcoxon test after multiple outputation — [p-value comment as in outcome 6, analysis 1]; Median Difference (Final Values) = 5, 95% CI 2-sided [-15 to 26] — Bootstrap

8. Secondary Outcome: Number of Participants Who Experienced Air Leaks
Description: Any pulmonary air leak (pulmonary interstitial emphysema, pneumothorax, pneumomediastinum) confirmed by chest x-ray
Time Frame: Participants will be followed for the duration of hospital stay, an expected average of 10 weeks
Population: The participants who had air leak at baseline (prior to randomization) were excluded from analysis (3 placebo and 5 azithromycin).
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (5% Dextrose) | Azithromycin
Number analyzed (Participants) | 57 | 55
Participants | 4 | 7
Statistical Analysis 1: Comparison: Placebo (5% Dextrose) vs Azithromycin; Test type: Superiority; p = 0.49, Fisher Exact

9. Secondary Outcome: Number of Participants Who Received Postnatal Steroids
Description: Receipt of steroid medications (hydrocortisone, dexamethasone)
Time Frame: 36 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (5% Dextrose) | Azithromycin
Number analyzed (Participants) | 61 | 60
Participants | 14 | 15
Statistical Analysis 1: Comparison: Placebo (5% Dextrose) vs Azithromycin; Test type: Superiority; p = 0.88, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.07, 95% CI 2-sided [0.44 to 2.63]

10. Secondary Outcome: Number of Participants Who Received Non-Study Antibiotics
Description: Received Non-study antibiotics following study drug intervention period.
Time Frame: Participants will be followed for the duration of hospital stay, an expected average of 10 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (5% Dextrose) | Azithromycin
Number analyzed (Participants) | 61 | 60
Participants | 14 | 8
Statistical Analysis 1: Comparison: Placebo (5% Dextrose) vs Azithromycin; Test type: Superiority; p = 0.18, Generalized Estimating Equations

11. Secondary Outcome: Pharmacokinetics (PK)/Pharmacodynamics (PD) Modelling of Time Course of Azithromycin Plasma Concentrations
Description: Number of serum azithromycin concentrations that fell outside the 90% prediction interval determined by 200 simulated replicates based on the population PK of azithromycin in preterm infants.
Time Frame: Study day 1-day 7
Population: No plasma samples from placebo group were analyzed for azithromycin concentrations
Measure: Number; unit: serum conc outside predicted interval
Units Other Than Participants: number of serum samples concentrations
Arm/Group | Placebo (5% Dextrose) | Azithromycin
Number analyzed (Participants) | 0 | 15
Number analyzed (number of serum samples concentrations) | 0 | 27
serum conc outside predicted interval |  | 4

12. Other Pre Specified Outcome: Number of Participants With Threshold Retinopathy of Prematurity (ROP)
Description: Threshold ROP requiring surgical intervention as diagnosed by ophthalmologic examination
Time Frame: Participants will be followed for the duration of hospital stay, an expected average of 10 weeks
Population: The number of participants who survived to receive at least 1 eye exam for retinopathy of prematurity
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (5% Dextrose) | Azithromycin
Number analyzed (Participants) | 56 | 56
Participants | 4 | 11
Statistical Analysis 1: Comparison: Placebo (5% Dextrose) vs Azithromycin; Test type: Superiority; p = 0.05, Generalized Estimating Equation

13. Other Pre Specified Outcome: Number of Participants With Necrotizing Enterocolitis (NEC)
Description: Necrotizing enterocolitis ≥ Bell Stage II by radiographic and clinical criteria.
Time Frame: Participants will be followed for the duration of hospital stay, an expected average of 10 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (5% Dextrose) | Azithromycin
Number analyzed (Participants) | 61 | 60
Participants | 5 | 4
Statistical Analysis 1: Comparison: Placebo (5% Dextrose) vs Azithromycin; Test type: Superiority; p = 1.0, Fisher Exact

14. Other Pre Specified Outcome: Number of Participants With Infections During the NICU Hospitalization
Description: Culture-confirmed bacterial or fungal infection based on culture from sterile site (blood, cerebral spinal fluid, or urine)
Time Frame: Participants will be followed for the duration of hospital stay, an expected average of 10 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (5% Dextrose) | Azithromycin
Number analyzed (Participants) | 61 | 60
Participants | 14 | 8
Statistical Analysis 1: Comparison: Placebo (5% Dextrose) vs Azithromycin; Test type: Superiority; p = 0.18, Generalized Estimating Equations

15. Other Pre Specified Outcome: Number of Participants With Severe Intraventicular Hemorrhage (IVH)
Description: Number of Participants with Grade III or IV IVH confirmed by cranial ultrasound
Time Frame: Participants will be followed for the duration of hospital stay, an expected average of 10 weeks
Population: The participants who had a Grade III or IV IVH at baseline (prior to randomization) were excluded (2 placebo and 4 Azithromycin).
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (5% Dextrose) | Azithromycin
Number analyzed (Participants) | 59 | 56
Participants | 2 | 7
Statistical Analysis 1: Comparison: Placebo (5% Dextrose) vs Azithromycin; Test type: Superiority; p = 0.091, Fisher Exact

16. Other Pre Specified Outcome: Number of Participants With Periventricular Leukomalacia (PVL)
Description: The number of Participants with cranial ultrasound confirmed PVL
Time Frame: Participants will be followed for the duration of hospital stay, an expected average of 10 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (5% Dextrose) | Azithromycin
Number analyzed (Participants) | 61 | 60
Participants | 5 | 4
Statistical Analysis 1: Comparison: Placebo (5% Dextrose) vs Azithromycin; Test type: Superiority; p = 1.0, Fisher Exact

17. Other Pre Specified Outcome: Number of Participants With Patent Ductus Arteriosus (PDA)
Description: Detection of PDA by cardiac echocardiogram with left to right shunting, or clinical evidence of murmur, bounding pulses, and widened pulse pressure.
Time Frame: 14 days
Population: Participants who did not have PDA at baseline (prior to randomization). Participants with PDA at baseline were excluded from analysis (5 placebo and 5 azithromycin.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (5% Dextrose) | Azithromycin
Number analyzed (Participants) | 56 | 55
Participants | 21 | 25
Statistical Analysis 1: Comparison: Placebo (5% Dextrose) vs Azithromycin; Test type: Superiority; p = 0.33, Generalized Estimating Equations

18. Other Pre Specified Outcome: Number of Participants With Cardiac Arrhythmia
Description: Number of Participants with EKG evidence of prolonged QT (QTc > 450 ms)
Time Frame: 3 days
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (5% Dextrose) | Azithromycin
Number analyzed (Participants) | 61 | 60
Participants | 0 | 0
Statistical Analysis 1: Comparison: Placebo (5% Dextrose) vs Azithromycin; Test type: Superiority; p = 1.0, Fisher Exact

ADVERSE EVENTS:
Time Frame: 3 years 6 months
Arm/Group | Placebo (5% Dextrose) | Azithromycin
All-Cause Mortality (participants affected / at risk) | 6/61 | 5/60
Serious Adverse Events (participants affected / at risk) | 39/61 | 44/60
Other Adverse Events (participants affected / at risk) | 51/61 | 51/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Placebo (5% Dextrose) (N=61) | Azithromycin (N=60)
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 6 | 5
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Apnea (Respiratory, thoracic and mediastinal disorders) | 4 | 3 — Breathing pause > 20 seconds
Patent Ductus Arteriosus (Cardiac disorders) | 12 | 17 — Patent ductus arteriosus confirmed by cardiac echocardiography
Necrotizing enterocolitis (Gastrointestinal disorders) | 3 | 3 — Necrotizing enterocolitis Bell Stage ≥2
Intestinal Perforation (Gastrointestinal disorders) | 4 | 3
Ileal stricture (Gastrointestinal disorders) | 0 | 1
Cholestasis (Hepatobiliary disorders) | 5 | 5
Retinopathy of prematurity (Eye disorders) | 3/60 | 11/58 — Retinopathy of prematurity (ROP) >Stage 2
Anemia (Blood and lymphatic system disorders) | 6 | 5 — hematocrit <25
White blood cell count >40,000 cells/mm3 (Blood and lymphatic system disorders) | 4 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 2 — platelet count <50,000
Sepsis (Infections and infestations) | 9 | 6 — Positive culture from a sterile site (blood or spinal fluid)
Urinary tract infection (Infections and infestations) | 4 | 0
Blood Urea Nitrogen > 60 mg/dL (Metabolism and nutrition disorders) | 4 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 2 | 0 — Serum calcium level >12.2 mg/dL
Hypochloremia (Metabolism and nutrition disorders) | 0 | 1 — Serum chloride <80 mEq/L
Hypernatremia (Metabolism and nutrition disorders) | 2 | 1 — Serum sodium >155 mEq/L
Hypokalemia (Metabolism and nutrition disorders) | 0 | 2 — Serum potassium <2.4 mEq/L
Hyponatremia (Metabolism and nutrition disorders) | 1 | 1 — Serum sodium <121 mEq/L
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (5% Dextrose) (N=61) | Azithromycin (N=60)
IV site reaction (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1
Gastric residual >50% volume of feed (Gastrointestinal disorders) | 1 | 3
Abdominal Distension (Gastrointestinal disorders) | 2 | 3 — Abdominal girth increase > 2cm from baseline
Loose stools (Gastrointestinal disorders) | 1 | 0 — stool consistency change with more water content <48 h duration
Oral thrush (Infections and infestations) | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 12 | 11 — white blood cell count >20,000 and <40,000 cells/mm3
Thrombocytopenia (Blood and lymphatic system disorders) | 12 | 4 — platelet count <100,000 and >50,000 cells/mm3
Abnormal liver function test (Hepatobiliary disorders) | 0 | 1 — Serum liver function test (AST/ALT/ or alkaline phosphatase) 1.5-3.5X normal value
conjugated hyperbilirubinemia (Hepatobiliary disorders) | 14 | 8 — Direct bilirubin 1.0-2.0 mg/dL
Elevated serum creatinine (Renal and urinary disorders) | 1 | 2 — Serum creatinine 1.3-2.3 mg/dL
Anemia (Blood and lymphatic system disorders) | 16 | 12 — hematocrit <35% and >25%
metabolic acidosis (Metabolism and nutrition disorders) | 18 | 19 — Serum bicarbonate <22 and >14 mEq/L
Metabolic alkalosis (Metabolism and nutrition disorders) | 6 | 8 — Serum bicarbonate >30 and <46 mEq/L
Elevated Blood Urea Nitrogen (Metabolism and nutrition disorders) | 28 | 26 — Serum BUN >27 and <60 mg/dL
Hyperkalemia (Metabolism and nutrition disorders) | 21 | 20 — Serum potassium >5.5 and <6.9 mEq/L
Hyperbilirubinemia (Hepatobiliary disorders) | 7 | 9 — Total bilirubin > 7 and <14 mg/dL
Hypernatremia (Metabolism and nutrition disorders) | 8 | 13 — Serum sodium <132 and >120 mEq/dL

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-01-30): https://cdn.clinicaltrials.gov/large-docs/34/NCT01778634/Prot_SAP_000.pdf
  • Informed Consent Form (2017-01-30): https://cdn.clinicaltrials.gov/large-docs/34/NCT01778634/ICF_001.pdf